CLINICAL TRIAL: NCT02991209
Title: A Randomized Double-blind Study of Testosterone Replacement Therapy or Placebo in Testicular Cancer Survivors With Mild Leydig Cell Insufficiency (Einstein-intervention)
Brief Title: Study of Testosterone vs Placebo in Testicular Cancer Survivors
Acronym: Einstein
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mikkel Bandak (Other)
Responsible Party: Sponsor-Investigator, Mikkel Bandak, MD, Research Fellow, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 010815Testis
Record Dates: First submitted 2016-11-25; First posted 2016-12-13 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Metabolic Syndrome; Testicular Cancer; Leydig Cell Failure in Adult
MeSH Terms: conditions — Metabolic Syndrome; Testicular Neoplasms | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tostran 2% (Experimental): 1 years treatment with transdermal Tostran 2%
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): 1 years treatment with placebo gel
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Testosterone
  Other Names: Tostran
  Arms: Tostran 2%
Drug: Placebos
  Arms: Placebo

SUMMARY:
The overall purpose of the study is to evaluate the effect of 12 months testosterone replacement therapy in testicular cancer survivors with mild Leydig Cell Insufficiency in order to reduce the risk of cardiovascular disease.

The primary study objective is to evaluate changes in insulin sensitivity. The secondary study objective is to evaluate changes in the prevalence of metabolic syndrome, body composition, systemic inflammation and symptoms of testosterone deficiency.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled intervention study, designed to evaluate the effect of testosterone replacement therapy in testicular cancer survivors with mild Leydig Cell Insufficiency.

70 subjects will be randomized to receive either testosterone replacement therapy or placebo. The subjects will be invited for an information meeting where informed consent is signed. If a subject is suitable for participation in the trial, subject will be randomized to testosterone replacement therapy or placebo and baseline investigations will be performed. Afterwards, a 52-weeks treatment period begins in which subjects receive a daily dose of testosterone or placebo. Dose adjustment will be made three times during the first 8 weeks of the study. Evaluation of primary and secondary endpoints will be performed after 26 weeks, at the end of treatment (52 weeks) and three months after completion of treatment (week 64).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Previous treatment for testicular cancer.
* No signs of relapse 1 year after last treatment (orchiectomy, radiotherapy, chemotherapy).
* Free testosterone < the age-adjusted median and > -2 standard deviations (SD) from the age-adjusted median and LH > 2 SD from the age-adjusted median.

Exclusion Criteria:

* Treatment with testosterone within the last 6 months.
* Contraindications to testosterone treatment (prostate cancer, prostate specific antigen (PSA)> 4 ng/mL), malignancy suspect prostate by digital rectal examination, Alanine aminotransferase (ALT)> 1.5 upper reference level, Erythrocyte Volume Fraction (EVF) > 50%.
* Breast cancer.
* Symptomatic obstructive sleep apnoea syndrome
* Heart failure > NYHA II.
* Uncontrolled hypertension: (Systolic blood pressure > 160 mm Hg despite antihypertensive treatment, measured at two separate occasions)
* Inability to understand information about the trial
* Participation in any other clinical trial
* Allergy for the active substance or additives in Tostran or placebo.
* Known diabetes mellitus, or diabetes mellitus detected at screening or baseline tests.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-11; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Changes in insulin sensitivity | 1 year
  Evaluation of changes in two hours plasma glucose investigated by Oral Glucose Tolerance Test (OGTT)

SECONDARY OUTCOMES:
Changes in fasting plasma lipids between baseline and 52 weeks | 1 year
Changes in BMD and fat percent between baseline 52 weeks | 1 year
  BMD and body composition evaluated by DXA-scan
Changes in systemic inflammation between baseline and 52 weeks | 1 year
  Analysis of tnf-alfa, interleukine 1-beta, interleukine 1, interleukine 6, interleukine 8
Changes in plasma-adipocytokines between baseline and 52 weeks | 1 year
Changes in fasting plasma glucose between baseline and 52 weeks | 1 year
Changes in Quality of life between baseline and 52 weeks. | 1 year
  EORTC-QLQ C30
Adverse events evaluated by the Common Terminology Criteria for Adverse Events Version 4.0 | 1 year
Changes in prevalence of metabolic syndrome between baseline and 52 weeks | 1 year
  According to NCEP-ATPIII criteria
Changes in haemoglobin A1c between baseline and 52 weeks | 1 year
Changes in plasma insulin between baseline and 52 weeks | 1 year
Changes in fatigue between baseline and 52 weeks | 1 year
  MFI-20 (Multidimensional Fatigue Inventory)
Changes in Anxiety and depression between baseline and 52 weeks | 1 year
  HADS (Hospital Anxiety and Depression Scale)
Changes in Symptoms of low levels of testosterone, erectile dysfunction between baseline and 52 weeks | 1 year
  IIEF-15 (International Index of Erectile Dysfunction)

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreiberg M, Jorgensen N, Juul A, Lauritsen J, Oturai P, Helge JW, Christensen JF, Aksglaede L, Schauer T, Wagner T, Rosenvilde J, Grunwald E, Dehlendorff C, Daugaard G, Bandak M. A randomized double-blind single center study of testosterone replacement therapy or placebo in testicular cancer survivors with mild Leydig cell insufficiency (Einstein-intervention). Clin Genitourin Cancer. 2022 Oct;20(5):404-414. doi: 10.1016/j.clgc.2022.04.017. Epub 2022 May 2. PMID 35701334
- [Derived] Hojer EG, Kreiberg M, Dehlendorff C, Jorgensen N, Juul A, Lauritsen J, Wagner T, Rosenvilde J, Daugaard G, Bandak M. Effect of Testosterone Replacement Therapy on Quality of Life and Sexual Function in Testicular Cancer Survivors With Mild Leydig Cell Insufficiency: Results From a Randomized Double-blind Trial. Clin Genitourin Cancer. 2022 Aug;20(4):334-343. doi: 10.1016/j.clgc.2022.03.012. Epub 2022 Apr 1. PMID 35514022
- [Derived] Priskorn L, Kreiberg M, Bandak M, Lauritsen J, Daugaard G, Petersen JH, Aksglaede L, Juul A, Jorgensen N. Testicular cancer survivors have shorter anogenital distance that is not increased by 1 year of testosterone replacement therapy. Hum Reprod. 2021 Aug 18;36(9):2443-2451. doi: 10.1093/humrep/deab162. PMID 34223605
- [Derived] Bandak M, Jorgensen N, Juul A, Lauritsen J, Kreiberg M, Oturai PS, Helge JW, Daugaard G. A randomized double-blind study of testosterone replacement therapy or placebo in testicular cancer survivors with mild Leydig cell insufficiency (Einstein-intervention). BMC Cancer. 2017 Jul 3;17(1):461. doi: 10.1186/s12885-017-3456-5. PMID 28673265